CLINICAL TRIAL: NCT02140632
Title: Local Steroid Injection vs Wrist Splinting for Carpal Tunnel Syndrome: A Randomized Clinical Trial
Brief Title: Efficacy Study of Local Steroid Injection and Wrist Splinting for Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Ho SO, Resident specialist, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR-13-018(64-16)
Record Dates: First submitted 2014-05-10; First posted 2014-05-16 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Carpal Tunnel Syndrome; Local Steroid Injection; Wrist Splinting
Keywords: Carpal tunnel syndrome; Local steroid injection; Wrist splinting
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local steroid injection (Experimental): The local injection of steroid is performed by the same investigator after the randomization. Using a sterile technique, 20mg methylprednisolone acetate premixed with lidnocaine is injected using a 25-gauge x 5/8" needle. The needle is inserted medially to the palmaris longus tendon at the distal palmar crease in the wrist at an angle of 45-degree to the forearm. The steroid is injected at approximately 1cm below the skin. The needle will be repositioned if there is any resistance to injection, or any pain or paraesthesia in the median nerve territory.
  Interventions: Procedure: Local methylprednisolone acetate and lidnocaine injection
- Wrist splinting (Active Comparator): After randomization, the hands of the patients in the splinting group are splinted in neutral position with standard cotton-polyester splint. Patients are encouraged to use the splints during nighttime whenever possible for one month.
  Interventions: Device: wrist splinting

INTERVENTIONS:
Procedure: Local methylprednisolone acetate and lidnocaine injection
  Other Names: depomedrol with lidnocaine
  Arms: Local steroid injection
Device: wrist splinting
  Arms: Wrist splinting

SUMMARY:
Carpal tunnel syndrome is caused by the compression of median nerve at the wrist where it passes through a narrow space called carpal tunnel formed by the wrist bones, ligaments and tendons. The common symptoms include numbness and pain over the areas supplied by the median nerve namely the thumb, the index finger, the middle finger and the outer part of the ring finger. There can be loss of sensation, weakness or muscle atrophy in severe cases. The functions of the affected hands may be greatly impaired.

Carpal tunnel syndrome is very common. It can lead to significant economic impact both to the affected individual and the society either by the direct treatment cost and indirectly from the working ability loss. Despite the vast burden, there is no consensus regarding its treatment so far. Surgery is generally effective and often reserved for severe cases. There are many nonsurgical treatment options. Local steroid injection and wrist splinting are among the commonest and with more evidence. Local steroid injection into the carpal tunnel can reduce the inflammation and swelling. Wrist splinting can maintain the wrist at its neutral position where the pressure at the carpal tunnel is the least. However, there are only very few studies comparing these two treatments directly.

Patients complaining of finger numbness who have been confirmed to have carpal tunnel syndrome by nerve conduction test are invited to participate in the study. The patients who agreed to be recruited are asked about their basic informations and the details of the carpal tunnel syndrome symptoms. Their hands will be examined. They are asked to fill in a questionnaire specific for assessing the symptom severity and the functional status of patients with carpal tunnel syndrome. They will then be assigned to one of the two treatment groups randomly and receive the respective treatment. They need to come back for follow-up at one month and to fill in the questionnaire again.

The study hypothesis is local steroid injection is more effective than wrist splinting in treating carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is caused by the pressure and consequent compression on the median nerve within a confined anatomical area at the wrist referred to as the carpal tunnel. It is very common and has an important socio-economic impact. The prevalence of CTS in the UK is 7-16%. Its incidence has been estimated at 88-125 per 100,000 in USA. Economic consequences include the direct financial implications of treatment and the indirect cost of absenteeism from the workplace. The median number of days away from work for CTS is among the highest at 27 days. In the US in 1995, between 400,000 and 500,000 patients underwent surgical decompression. This equates to an economic cost of in excess of $2 billion. CTS and hearing loss was found to account for more morbidity, measured by cases and working days lost, than any other illness in the US working population. CTS may also occur as a work- related disorder leading to compensation claims.

Despite the vast burden of the disease, there is no consensus regarding its best management. Surgical treatment is generally preferred in severe cases of CTS. A Cochrane review investigating surgical treatment of CTS showed surgical treatment relieves symptoms significantly better than splinting, but no conclusion could be drawn in people with mild symptoms and if surgical treatment is better than steroid injection. On the other hand, surgical treatment is relatively costly and carries risks of significant complications that may last several months and give rise to further work absence. In addition, the waiting time for surgery is usually long.

For non-surgical interventions many modalities have been trialed but only a few have shown discernable benefits. Local steroid injection and wrist splinting are among the most popular options. They are commonly employed in mild to moderate cases of CTS. For severe cases, they can also offer relief of complaints during the waiting period for surgery or when there are contra-indications for surgery. Systematic reviews of randomized controlled trials have concluded that local steroid injection provides greater clinical improvement at one month compared with placebo and that there is weak evidence that a splint worn at night is more effective than no treatment in the short term. However, the number of studies that compare the two methods is limited, and they are mostly either retrospective in design or prospective but non-randomized. Two randomized controlled trials comparing local steroid injection and splinting found respectively that local steroid injection does not significantly improve clinical outcome compared to anti-inflammatory drugs and splinting and that injections of steroids are ineffective. However, the conclusions of these two studies are limited either by a small sample size or the lack of a validated outcome measure.

We would like to conduct a prospective randomized clinical trial comparing the efficacy of local steroid injection and splinting in patients with CTS using the Boston Carpal Tunnel Questionnaire as outcome measure with a 4-week follow-up.

Patients attending the medical clinic of a local hospital (Kwong Wah Hospital) complaining of finger or hand numbness are referred to the electro-neuro-diagnostic unit for nerve conduction test. Consecutive patients with clinical and electrophysiological features of CTS are invited to participate in the study. Clinical features are pain, paresthesia or weakness in the median nerve distribution for at least 3 months. The neurodiagnostic criteria are based on the American Academy of Neurology summary statement, which further classifies the abnormalities as follows: (1) mild abnormality, i.e., abnormal comparative tests or prolonged median distal sensory latency (DSL > 3.5 ms) but normal median distal motor latency (DML); (2) moderate abnormality, i.e., prolonged median DSL and DML (⩾4.2 ms); and (3) severe abnormality, i.e., absence of median sensory nerve action potential and prolonged median DML or absent compound muscle action potentials.

Patients are excluded if they have any recognized causes of CTS including inflammatory arthritis, diabetes mellitus, hypothyroidism, renal failure, polyneuropathy and history of significant local trauma. Other exclusion criteria include age younger than 18 years, previous treatment of CTS and pregnancy. Patients with motor impairment or thenar muscle atrophy are also excluded and they will be referred to the Orthopedic unit for assessment of surgery.

All potential participants are informed of the objectives and procedures of this study, as well as the possible complications. The patients who have given informed consent are interviewed by a single investigator within 4 weeks of the NCV. Their demographical data including age, gender and body mass index (BMI) are recorded. The duration of the symptoms, medical comorbidities and employment status are documented. Examination of the hand is performed by the same investigator focusing on the sensory loss at the tips of digits 1, 2, 3, or the medial side of digit 4, and weakness or atrophy of the abductor pollicis brevis or opponens pollicis. Sensation is assessed using pinpricks. Sensory and motor function is recorded to be either normal or impaired. In patients with bilateral CTS, the most symptomatic hand will be included. In case both hands are equally symptomatic, the dominant hand will be included. Recruited patients are asked to complete the Boston Carpal Tunnel Questionnaire (BCTQ). They will then be allocated to one of the two treatment arms according to the randomization procedure.

Patients are randomly assigned to one of the two treatment groups using sequentially numbered opaque sealed envelopes (SNOSE). Allocation concealment is maintained before the randomization procedure.

The local injection of steroid is performed by the same investigator after the randomization. Using a sterile technique, 20mg depomedrol premixed with lidnocaine is injected using a 25-gauge x 5/8" needle. The needle is inserted medially to the palmaris longus tendon at the distal palmar crease in the wrist at an angle of 45-degree to the forearm. The steroid is injected at approximately 1cm below the skin. The needle will be repositioned if there is any resistance to injection, or any pain or paraesthesia in the median nerve territory.

Minor complications of steroid injection include local pain, bleeding, skin depigmentation, skin atrophy and digital ischemia. Concerns that nerve or tendon injury may result from steroid injection appear to be unfounded. In 28 studies of local steroid injection treatment involving 1981 hands in total there have been no reported instances of such injury, suggesting that the risk is very low. There is a small risk of infection.

After randomization, the hands of the patients in the splinting group are splinted in neutral position with standard cotton-polyester splint. Patients are encouraged to use the splints during nighttime whenever possible for 1 months.

The potential side effects of splinting include discomfort due to the local pressure and allergic response to the splint material.

The primary outcome measure is clinical improvement at one month. The Boston Carpal Tunnel Questionnaire (BCTQ) is used as the measure assessing clinical response. It is a self-administered disease-specific questionnaire for assessing severity of symptoms and functional status based on two scales. The symptom severity scale (SSS) is comprised of 11 questions, and the functional status scale (FSS) is comprised of 8 questions. The assessment of each question is on a scale of 1-5 points, in which 1 indicates no symptom, and 5 indicates severe symptoms. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5. The evidence base of the psychometric properties indicates that the BCTQ is a valid, reliable, responsive and acceptable instrument and should be included as a primary outcome measures in CTS intervention trials. The questionnaire has Chinese validity.

Patients are interviewed at one month after randomization. They are asked to complete the BCTQ and rate the satisfaction of treatment each time. Duration of sick leave for employed patients, concomitant use of analgesics, and adverse effects are recorded.

As all participants have symptoms of CTS and will receive valid active treatments, they should be motivated and compliant to the protocol. They are encouraged to report to the PI should there be any problems occurred regarding the splints or any adverse effects developed in both treatment groups. Appropriate actions will be taken or advices given by the PI. The subjects in the splinting group are instructed to mark each night that they have worn the splints on a calendar. Subjects who missed the scheduled follow-up will be contacted and encouraged to attend the re-scheduled follow-up as soon as possible.

Based on previous studies, the minimum clinically important difference is 0.74 for the BCTQ. With 90% statistical power, 5% significance level, and two-sided statistical tests, and assuming a standard deviation of 0.8 for the BCTQ score the study can detect a true difference of at least 0.74 point on the BCTQ between the two intervention groups when 50 patients are randomized. Version 20.0 of the SPSS statistical package is used. Descriptive statistics are presented as frequencies, means with standard deviation or medians with ranges as appropriate. Baseline parameters of patient between two treatment groups are compared by chi-square test for categorical variables, Student's t test for continuous variables with normal distribution or Mann-Whitney U test for nonparametric continuous variables. BCTQ scores before treatment and at the one, four and twelve weeks after treatment are compared with paired samples t test. Differences of the BCTQ scores between the two treatment groups were investigated with independent samples t test. For multi-variate analysis, multiple linear regression is used to compute the differences of outcome measures between the two treatment groups, and within the groups before and after the respective treatments with adjustment for baseline variables. Results are considered statistically significant if the P value is less than 0.05.

This trial has been approved by the local ethics committee (Kowloon West Cluster Ethical Committee). The trial will be conducted in full compliance with the Helsinki Declaration and the Guideline for Good Clinical Practice of the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use.

ELIGIBILITY:
Inclusion Criteria:

* patients attending the medical clinic of Kwong Wah Hospital with clinical and electrophysiological features of CTS

Exclusion Criteria:

* any recognized causes of CTS including inflammatory arthritis, diabetes mellitus, hypothyroidism, renal failure, polyneuropathy and history of significant local trauma
* previous treatment of CTS
* pregnancy
* patients with motor impairment or thenar muscle atrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical improvement at one month | One month after treatment
  The Boston Carpal Tunnel Questionnaire is used as the measure assessing clinical response. It is a self-administered disease-specific questionnaire for assessing severity of symptoms and functional status based on two scales. The symptom severity scale is comprised of 11 questions, and the functional status scale is comprised of 8 questions. The assessment of each question is on a scale of 1-5 points, in which 1 indicates no symptom, and 5 indicates severe symptoms. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5.

SECONDARY OUTCOMES:
Patient satisfaction at one month | One month after treatment
  Assessment of patient satisfaction is classified on a 5-point scale as completely satisfied, almost satisfied, moderately satisfied, somewhat satisfied, and dissatisfied.
Side effects | One month after treatment
  Any side effects thought to be related to the interventions are documented.
Prognostic factor - Age | One month after treatment
  The association between age and the response to treatment (symptom severity scale and functional status scale) is assessed.
Prognostic factor - Gender | One month after treatment
  The association between gender and the response to treatment (symptom severity scale and functional status scale) is assessed.
Prognostic factor - Duration of symptoms | One month after treatment
  The association between the duration of symptoms and the response to treatment (symptom severity scale and functional status scale) is assessed.
Prognostic factor - Presence or absence of sensory deficit | One month after treatment
  The association between the presence or absence of sensory deficit and the response to treatment (symptom severity scale and functional status scale) is assessed.
Prognostic factor - Nerve conduction velocity severity | One month after treatment
  The association between the nerve conduction velocity severity (1-3) and the response to treatment (symptom severity scale and functional status scale) is assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ho So, MBBS, Principal Investigator — Kwong Wah Hospital
Locations (1):
- Kwong Wah Hospital, Kowloon, Hong Kong, China